CLINICAL TRIAL: NCT00000590
Title: Anti-HIV Immunoglobulin (HIVIG) in Prevention of Maternal-Fetal HIV Transmission (Pediatric ACTG Protocol 185)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 310
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2005-03

CONDITIONS: Acquired Immunodeficiency Syndrome; Disease Transmission, Vertical; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Immunoglobulins

INTERVENTIONS:
Drug: immunoglobulins

SUMMARY:
To determine if HIV hyperimmune globulin (HIVIG) given to HIV-positive pregnant women during the second and third trimester of pregnancy reduced the likelihood of maternal-fetal HIV transmission. Conducted in collaboration with the National Institute of Child Health and Human Development and the National Institute of Allergy and Infectious Diseases. The trial was Pediatric ACTG Protocol 185.

DETAILED DESCRIPTION:
BACKGROUND:

The HIV epidemic in the United States has changed its course in the past few years. The main risk group of the past, homosexual males, has reduced numbers of new infections because of education and prevention. Other groups, including intravenous drug abusers, disadvantaged urban socioeconomic classes and adolescents, continue to be infected and to transmit HIV by needle sharing and/or unprotected heterosexual activity. Many of these newly infected individuals are women of child-bearing age. These women in turn infect their children. The Centers for Disease Control estimates that there will be 2,000 infected infants born to 6,000 HIV-positive mothers annually in the United States.

Over the past few years, several studies have identified the risk of maternal-fetal transmission of HIV by seropositive mothers. The risk is close to 30 percent. However, for reasons not yet understood, the risk appears to be higher in Africa, approaching 40 percent, and lower in Europe, approaching 16 percent. Factors influencing maternal-fetal transmission of HIV are not well defined but may include the clinical state of the mother, plasma p24 antigen positivity of the mother, viral load, prior pregnancy associated with maternal-fetal HIV transmission, absence of maternal epitope specific and/or high affinity gp120 antibodies, or prematurity.

The results of a Phase III, multicenter, double-blind, randomized, placebo-controlled clinical trial to evaluate the efficacy, safety, and tolerance of zidovudine for the prevention of HIV transmission from infected pregnant women to their infants (ACTG protocol 076) provided for the first time proof of the concept that a preventive intervention can reduce vertical HIV transmission (47). Based on analysis of data for 364 evaluable births, zidovudine (ZDV or AZT) treatment according to the regimen employed in ACTG 076 appeared to reduce the risk of HIV transmission by two thirds, from 25.5 percent to 8.3 percent. Eligible subjects were HIV-infected pregnant women who had received no antiretroviral therapy during their current pregnancy, who had no maternal clinical indications for antiretroviral therapy, and who had CD4+ T-lymphocyte counts above 200 per microliter at study entry.

Efficacy of ZDV for reduction of vertical HIV transmission in women with advanced HIV disease who are already receiving antiretroviral treatment according to current clinical indications for their own health, or with CD4+ T-lymphocyte counts of 200 per microliter or below, or both was not evaluated in ACTG 076.

Administration of an antiretroviral agent to a pregnant woman in theory could reduce the risk of neonatal infection by reducing the exposure of the fetus to maternal virus, or by prophylaxis of the fetus prior to exposure. Because it is postulated that intense exposure of a potentially uninfected fetus to HIV present in maternal blood and genital tract secretions occurs during parturition, the design of this study includes intrapartum administration of ZDV followed by six weeks of oral ZDV to the infant.

An identical regimen for ZDV administration was employed in ACTG Protocol 076.

Pediatric ACTG Protocol 185 evaluated the hypothesis that in HIV-infected pregnant women receiving oral ZDV for medical indications, HIVIG administered monthly beginning at 20-30 weeks gestation in combination with intravenous ZDV intrapartum, together with a single newborn dose of HIVIG within 12 hours after birth in combination with six weeks of newborn oral ZDV, would reduce vertical HIV transmission compared with IVIG administered identically as a control agent.

DESIGN NARRATIVE:

Randomized, double-blind, controlled. Approximately half of the women were given intravenous HIVIG every four weeks until delivery. The other half received standard intravenous immunoglobulin (IVIG) without anti-HIV antibody. Both groups received AZT. A similar dose of HIVIG or IVIG was given to the newborn infant within 12 hours of birth. Each infant of a multiple birth received the mother's randomized study drug. Infant blood samples were taken at birth and at several intervals during the first 24 months of life to determine the infants' HIV status by p24 antigen assays, plasma viremia, or HIV co-culture assays. An existing NICHD contract with Westat, Inc. was used to conduct the trial. Westat, the study coordinating center subcontracted to 25 NICHD clinical trial units. An approximately similar number of NIAID clinical trial units also participated in the trial. As of February 1, 1996, there were 51 clinical trial units participating. Data analysis was performed by Westat. In 1993, NHLBI contracted with North American Biologics to supply HIVIG. The trial ended in December, 1996.

ELIGIBILITY:
HIV-positive, asymptomatic, pregnant women with CD4 concentrations of 500 or less and their infants.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1991-09; Study Completion 1996-12

CONTACTS AND LOCATIONS:
Overall Officials: Steven Durako — Westat, Inc

REFERENCES:
- [Background] Lambert JS, Mofenson LM, Fletcher CV, Moye J Jr, Stiehm ER, Meyer WA 3rd, Nemo GJ, Mathieson BJ, Hirsch G, Sapan CV, Cummins LM, Jimenez E, O'Neill E, Kovacs A, Stek A. Safety and pharmacokinetics of hyperimmune anti-human immunodeficiency virus (HIV) immunoglobulin administered to HIV-infected pregnant women and their newborns. Pediatric AIDS Clinical Trials Group Protocol 185 Pharmacokinetic Study Group. J Infect Dis. 1997 Feb;175(2):283-91. doi: 10.1093/infdis/175.2.283. PMID 9203648
- [Background] Mofenson LM, Lambert JS, Stiehm ER, Bethel J, Meyer WA 3rd, Whitehouse J, Moye J Jr, Reichelderfer P, Harris DR, Fowler MG, Mathieson BJ, Nemo GJ. Risk factors for perinatal transmission of human immunodeficiency virus type 1 in women treated with zidovudine. Pediatric AIDS Clinical Trials Group Study 185 Team. N Engl J Med. 1999 Aug 5;341(6):385-93. doi: 10.1056/NEJM199908053410601. PMID 10432323
- Available data/document: Individual Participant Data Set: PACTG — http://biolincc.nhlbi.nih.gov/studies/pactg/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/pactg/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/pactg/